CLINICAL TRIAL: NCT00167726
Title: Neuraxial and Neurolytic Analgesia for Intractable Pain
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0482
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect longitudinal data on outcomes of neuraxial or neurolytic procedures in patients with intractable cancer and chronic noncancer pain so that we may contribute to the growing evidence for or against these therapies and to provide data for ongoing quality improvement activities.

ELIGIBILITY:
Inclusion Criteria:

* treated for intractable pain by the UW Interventional Pain Treatment program
* inpatient or outpatient

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective case series analysis. Subjects over the age of 18 who are offered neuraxial (epidural or intrathecal) analgesia or neurolytic procedures (e.g. celiac, hypogastric, or sacral nerve plexus block) to treat intractable pain through the UW Interventional Pain Program.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2005-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Prospective review of pain | six years
  The purpose of this study was to collect longitudinal data on outcomes of neuraxial or neurolytic procedures in patients with intractable cancer and chronic noncancer pain so that we may contribute to the growing evidence for or against these therapies and to provide data for ongoing quality improvement activities.

CONTACTS AND LOCATIONS:
Overall Officials: Nalini Sehgal, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States